CLINICAL TRIAL: NCT04943887
Title: Clinical Trial of a Telehealth Group-Based Intervention to Improve Mood in Underrepresented Individuals With Multiple Sclerosis: The Connect Trial (CONNECT)
Brief Title: CONNECT Trial of eSupport Online Health-coach Moderated Support Groups for Multiple Sclerosis
Acronym: CONNECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: eSupport Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MSO01-P001
Record Dates: First submitted 2021-06-14; First posted 2021-06-29 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Multiple Sclerosis
Keywords: Online Support Group
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Each participant will serve as his/her own control; after a 12-week waitlist control period, each participant will complete a 12-week treatment period [note that the very first group of enrolled participants (N ~10) will not have a waitlist period, but will instead enter directly into the 12-week treatment period].
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PwMS eSupport Groups (Experimental): 12-weeks active treatment of eSupport Health's Weekly Group Sessions, a formal semi-structured program of psychoeducational support delivered in a small group format by licensed therapists who specialize in MS. The active treatment period will follow a 12-week waitlist period that will be used to enable a within-subject control design. Note that the very first group enrolled (N~10) will not have a 12-week waitlist period but will instead enter directly into the 12-week treatment.
  Interventions: Behavioral: eSupport Health Weekly Group Sessions for PwMS

INTERVENTIONS:
Behavioral: eSupport Health Weekly Group Sessions for PwMS — A formal semi-structured program of psychoeducational support delivered in an online weekly small group format by health coaches (licensed therapists) who specialize in MS.

SUMMARY:
Within-subject waitlist-control group design trial of eSupport health-coach moderated online support group participation to address mental health needs in persons with multiple sclerosis (PwMS) from historically underrepresented groups (i.e., Black and Latinx patients).

DETAILED DESCRIPTION:
The purpose of this research is to see how well a new online eSupport Health Weekly Group Sessions program addresses the needs and improves the mood of adults with MS. This study is focusing on improving the online eSupport Weekly Group Session program for people with MS while assessing the impact of the program, particularly for Black and Latinx individuals as clinical research has often not included their experience.

The entire study is done remotely by computer, tablet, or smartphone with a web camera and with a stable internet connection. Subjects will be enrolled into closed, private, health-coach facilitated online support groups called eSupport Health Weekly Group Sessions. These sessions are hosted on eSupport Health's proprietary Zoom-based secure HIPAA-compliant telehealth platform. Each group is expected to have 10 participants and will meet weekly for 12 weeks. A licensed therapist ("Study Coach") leads the group sessions. The company's Mutual Respect & Trust (MRT)-based coaching method is utilized.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form (ICF)
* Able to speak, read and understand English
* Reside in the U.S.
* Willingness to enroll as a member in eSupport Health
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Willingness to adhere to the schedule of weekly online meetings with a minimum of 50% attendance (i.e., 6 of 12 meetings)
* Males and females; Age 18+
* Self-reported diagnosis of multiple sclerosis including the date of the diagnosis (month and year) and the name of the diagnosing physician
* Access to necessary resources for participating in a technology-based intervention (i.e., computer or tablet with a web camera and with a stable internet connection in a private setting) and demonstrated basic ability to use a computer by completing the electronic ICF completion process and meeting with the Study Coach via Zoom Telehealth secured platform at the Enrollment Session.
* Provide identification to verify name, date of birth, and address.

Exclusion Criteria:

1. Current participation in another treatment or intervention study
2. Presence of a condition(s) or diagnosis, either physical or psychological that precludes participation such as significant brain injury and developmental disability
3. Current suicidal intent
4. Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Adherence and completion | through study completion, 20-40 weeks
  The primary objective is to establish feasibility, defined as acceptable rates of <1> adherence, and <2> completion.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | through study completion, up to 40 weeks
  The primary efficacy outcome is to determine whether participation in 12-weeks of eSupport Health online groups results in decreased anxiety or depression.

OTHER OUTCOMES:
Functional Assessment in MS (FAMS) | through study completion, up to 40 weeks
  A tertiary objective is to determine efficacy: whether participation in 12-weeks of eSupport Health online groups results in improved quality of life.
UCLA Loneliness Scale Version 3 | through study completion, up to 40 weeks
  A tertiary objective is to determine efficacy: whether participation in 12-weeks of eSupport Health online groups results in decreased loneliness.
Treatment adherence / healthcare utilization | through study completion, up to 40 weeks
  A tertiary objective is to evaluate change in treatment adherence / healthcare utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria M Leavitt, Leavitt, Principal Investigator — eSupport Health, PBC
Locations (1):
- eSupport Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: CSR
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.